CLINICAL TRIAL: NCT05178342
Title: A Phase II, Open-Label, Multicenter Study of Orally Administered CA-4948 for the Treatment of Anemia in Patients With Very Low, Low or Intermediate Risk Myelodysplastic Syndromes (MDS)
Brief Title: Treatment of Anemia in Patients With Very Low, Low or Intermediate Risk Myelodysplastic Syndromes With CA-4948
Acronym: LUCAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Prematurely according to trial protocol
Sponsor: University of Leipzig (Other)
Collaborators: Curis, Inc. (Industry)
Responsible Party: Principal Investigator, Uwe Platzbecker, Prof. Dr., University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUCAS
Record Dates: First submitted 2021-11-02; First posted 2022-01-05 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Myelodysplastic Syndromes; Anemia
Keywords: MDS; Anemia; Myelodysplastic Syndrome; IRAK4
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — CA-4948

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CA-4948 treatment (Other): Single-arm design. all patients are treated with IMP
  Interventions: Drug: CA-4948

INTERVENTIONS:
Drug: CA-4948 — Patients will be treated orally with CA-4948 at 300 mg BID (2x200mg) over 4 cycles. One cycle consists of 28 days, 21 of which are treatment days, followed by 7 days off.
  Patients with erythroid response (HI-E) after 4 cycles who tolerate CA-4948 may continue to receive CA-4948 until loss of HI-E response.
  Other Names: Emavusertib

SUMMARY:
Anemia in LR-MDS patients

DETAILED DESCRIPTION:
Anemia in non-transfusion dependent (NTD) or transfusion dependent (low or high transfusion burden, LTB/HTB) patients with very low, low or intermediate risk myelodysplastic syndromes

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of de novo myelodysplastic syndrome (MDS) OR de novo myelodysplastic/myeloproliferative neoplasias (MDS/MPN) including MDS/MPN-RS-T, MDS/MPNu, aCML or CMML
2. Very low/low/intermediate risk disease: IPSS-R up to 3.5 for MDS; MDS/MPN < 10% bone marrow blasts; for CMML low or intermediate risk according to CPSS-Score
3. Symptomatic anemia (based on valid and complete hemoglobin and transfusion history):

   * NTD (non transfusion dependent): < 3 RBC transfusions and mean hemoglobin level <10 g/dl within the last 16 weeks
   * LTB (low transfusion burden): 3-7 RBC transfusions within the last 16 weeks in at least two transfusion episodes, maximum 3 in 8 weeks
   * HTB (high transfusion burden): ≥ 8 RBC transfusions within the last 16 weeks, ≥ 4 in 8 weeks
4. Defined transfusion strategy
5. No available option of an approved MDS therapy and classification of prior erythropoiesis-stimulating agent (ESA) treatment as follows:

   * Cohort A: ESA exposed (and refractory or intolerant)
   * Cohort B: ESA naive AND serum erythropoietin level >200 U/L

Exclusion Criteria:

Compliance with major study procedures

* Inability to swallow and retain oral medications (> 10 pills)
* Patient does not accept bone marrow sampling during screening and after the treatment
* Patient does not accept up to weekly peripheral blood sampling during screening and treatment

Safety

* ECOG performance status ≥ 3
* Inacceptable organ function

  1. Serum creatinine > 2 × ULN or calculated creatinine clearance < 30 ml/min
  2. AST > 2 × ULN or ALT > 2 × ULN
  3. total bilirubin > 2 × ULN (exception >3 × ULN in patients with documented Gilbert's syndrome)

Interfering treatments

* Prior treatment with azacitidine or decitabine
* Treatment with erythropoiesis stimulating agent (ESA), G-CSF, GM-CSF, lenalidomide, luspatercept and/or another investigational drug or device up to 14 days before registration
* Treatment with iron chelation therapy 56 days before registration, except for subjects on a stable or decreasing dose for at least eight weeks prior to inclusion and during study treatment
* Major surgery within 28 days prior to registration

Concomitant diseases

* Known human immunodeficiency virus infection (HIV)
* Active infectious hepatitis (HBV or HCV)
* Hepatitis virus detectable within 6 months before registration in patients with a history of hepatitis
* History of other invasive malignancy, unless definitively treated with curative intent, provided it is deemed to be at low risk for recurrence by the treating physician
* Presence of an acute or chronic toxicity resulting from prior anti-cancer therapy that has not resolved to Grade ≤ 1 (except anemia and alopecia)
* Known allergy or hypersensitivity to any component of the formulation of CA-494824
* Severe cardiovascular disease (e.g. myocardial infarction within 6 months registration, unstable angina within 6 months registration, NYHA Class III or greater congestive heart failure, serious arrhythmias uncontrolled on treatment, clinically significant pericardial disease, known QTc abnormality > 450 msec on ECG

Formal requirements

* Positive serum pregnancy test in women of childbearing potential
* Women of childbearing potential and men who partner with a woman of childbearing potential unwilling to use highly effective contraceptive methods for the duration of the study and for 90 days after the last dose of CA-4948
* Age under 18 years at registration
* Inability to provide written informed consent
* Simultaneous participation in another interventional clinical trial or participation in any clinical trial involving administration of an investigational medicinal product within 28 days prior registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Erythroid response (HI-E) | At the end of cycle 4 (each cycle is 28 days).
  To evaluate the proportion of patients who have an erythroid response (HI-E) according to the modified IWG 2018 criteria separately for both independent substudies.

SECONDARY OUTCOMES:
HI-E response (erythroid response) duration | From the date of treatment start until date of documented loss of response, assessed up to 30 months.
  To evaluate HI-E response from the first day of response until loss of response.
Time to HI-E (erythroid response) | From the date of treatment start until first day of response, assessed up to end of cycle 4 (each cycle is 28 days).
  To evaluate the time between start of treatment and first day of response.
Red blood cell (RBC) transfusions | From the date of treatment start until the date of end of treatment, assessed up to 30 months.
  To evaluate frequency of red blood cell transfusions in transfusion dependent patients
Neutrophil (HI-N) responses | At the end of cycle 4 (each cycle is 28 days).
  Neutrophil (HI-N) responses according to IWG 2018 criteria
Platelet (HI-P) responses | At the end of cycle 4 (each cycle is 28 days).
  Platelet (HI-P) responses according to IWG 2018 criteria
Safety of CA-4948 (toxicities and adverse events) | From the date of treatment start until the end of study, assessed up to 30 months.
  Assessments will include characterization of toxicities; characterization of AEs including type, incidence, severity, seriousness, and relationship to treatment
Number of participants with clinically significant changes of selected laborotory parameters (parameters listed in detailed description) | From the date of treatment start until the end of study, assessed up to 30 months.
  To ensure patient safety, close monitoring is carried and includes the analysis of: transaminases, bilirubin, amylase, lipase, troponin, lactate dehydrogenase, creatine kinase, uric acid, TSH, FT4, urine analysis.
Impact of treatment assessed by using the validated European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30) | From the date of treatment start until the end of study, assessed up to 30 months.
  To assess patient-reported quality of life during CA-4948 treatment: 30 questions assessing the quality of life of oncology patients across 10 subscales will be analyzed. All subscales have a score range from 0 to 100 points.
  Function subscales: a higher score represents a higher quality of life. Symptoms subscales: higher score represents higher level of symptoms/problems, i.e., represents lower quality of life.
Impact of treatment assessed by using the validated European Organisation for Research and Treatment of Cancer cancer related fatigue questionnaire (EORTC QLQ- FA12) | From the date of treatment start until the end of study, assessed up to 30 months.
  To assess patient-reported quality of life during CA-4948 treatment: 12 items, with four response categories for each item (coded with values from 1 to 4) will be analyzed. FA12 scores are transformed to the range 0-100: Higher levels indicate greater degrees of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof. Dr., Principal Investigator — University Leipzig
Locations (15):
- Germany (15):
  - Charité Berlin - Campus Benjamin Franklin, Med. Klinik m. S. Hämatologie, Onkologie, Tumorimmunologie, Berlin
  - Carl-Thiem-Klinikum Cottbus gGmbH, 2. Med. Klinik, Cottbus
  - Gemeinschaftspraxis Dr. Jacobasch Dresden, Hämatologie Onkologie, Dresden
  - Marienhospital Düsseldorf, Klinik für Onkologie und Hämatologie, Palliativmedizin, Düsseldorf
  - ONCOSEARCH, Institut für Klinische Studien GbR, Erlangen
  - InVO-Institut für Versorgungsforschung in der Onkologie, Koblenz
  - VK & K Studien GbR, Studienzentrum, Landshut
  - University Leipzig, Medizinische Klinik und Poliklinik I - Hämatologie und Zelltherapie, Hämostaseologie, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Klinik für Hämatologie und Onkologie Campus Lübeck, Lübeck
  - Universitätsklinikum Mainz, III. Medizinische Klinik und Poliklinik - Hämatologie, Internistische Onkologie und Pneumologie, Mainz
  - Universitätsklinikum Mannheim, III. Medizinische Klinik - Hämatologie und Onkologie, Mannheim
  - Klinikum Hochsauerland GmbH, Klinik f. Hämatologie, Onkologie, Palliativmedizin, Stammzelltransplantation, Meschede
  - Klinikum rechts der Isar der TU München III. Medizinische Klinik - Hämatologie und Onkologie, München
  - Friedrich-Ebert-Krankenhaus GmbH, Klinik für Hämatologie, Onkologie und Nephrologie, Neumünster
  - Rems-Murr-Kliniken gGmbH, Hämatologie, Onkologie und Palliativmedizin, Winnenden

IPD SHARING:
Plan to Share IPD: No